CLINICAL TRIAL: NCT00387309
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Intravenous Methylnaltrexone (MOA-728) for the Treatment of Post Operative Ileus.
Brief Title: Study Evaluating IV Methylnaltrexone for the Treatment of Post Operative Ileus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3200L2-300
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Post Operative Bowel Dysfunction
Keywords: Bowel
MeSH Terms: interventions — methylnaltrexone

INTERVENTIONS:
Drug: Methylnaltrexone (MOA-728)

SUMMARY:
Primary Objective: In subjects who have undergone segmental colectomy, the time between the end of surgery and first bowel movement is significantly shorter with the investigational MOA-728 regimen than with a placebo regimen.

ELIGIBILITY:
Inclusion:

* Must be scheduled for a segmental colectomy via open laparotomy with general anesthesia
* Subjects with history of inflammatory bowel disease are eligible as long as the disease is not currently active and all other criteria are met
* Subjects must meet the American Society of Anesthesiologists physical status I, II or III

Exclusion:

* Subjects who are scheduled for laparoscopic surgery for the segmental colectomy
* Subjects with a recent history (<1 year prior to randomization) of abdominal radiation therapy; Subjects with a history of small bowel obstruction, known or suspected bowel adhesions (other than minor, clinically nonsignificant adhesions)
* Subjects undergoing operations resulting in gastrointestinal ostomies, or who require use of post operative nonsteroidal anti-inflammatory drugs (NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495
Dates: Start 2006-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary Objective: In subjects who have undergone segmental colectomy, the time between the end of surgery and first bowel movement is significantly shorter with the MOA-728 regimen than with a placebo regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (82):
- United States (54):
  - Mobile, Alabama
  - Fort Smith, Arkansas
  - Chula Vista, California
  - Colton, California
  - Los Angeles, California
  - Oceanside, California
  - Palo Alto, California
  - San Jose, California
  - Torrance, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Bay Minette, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Naples, Florida
  - St. Petersburg, Florida
  - Vero Beach, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Naperville, Illinois
  - Park Ridge, Illinois
  - Kansas City, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Saint Paul, Minnesota
  - Albany, New York
  - Kingston, New York
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Danville, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Pawtucket, Rhode Island
  - Providence, Rhode Island
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Winchester, Virginia
- Australia (3):
  - Camperdown, New South Wales
  - Elizabeth Vale, South Australia
  - Woodville South, South Australia
- Germany (4):
  - Berlin
  - Halle
  - Heidelberg
  - München
- Hungary (4):
  - Budapest
  - Győr
  - Pécs
  - Székesfehérvár
- Italy (7):
  - Osio Sotto, Zingonia
  - Bologna
  - Ferrara
  - Genova
  - Monza
  - Padua
  - Roma
- Poland (4):
  - Katowice
  - Krakow
  - Lodz
  - Poznan
- Bucharest, Romania
- Beograd, Serbia and Montenegro
- South Africa (3):
  - Pretoria, Gauteng
  - Pietermaritzburg, KwaZulu-Natal
  - Cape Town, Western Cape
- Seoul, South Korea

REFERENCES:
- [Derived] Yu CS, Chun HK, Stambler N, Carpenito J, Schulman S, Tzanis E, Randazzo B. Safety and efficacy of methylnaltrexone in shortening the duration of postoperative ileus following segmental colectomy: results of two randomized, placebo-controlled phase 3 trials. Dis Colon Rectum. 2011 May;54(5):570-8. doi: 10.1007/DCR.0b013e3182092bde. PMID 21471758